CLINICAL TRIAL: NCT02467920
Title: Efficacy and Safety of Basal Insulin Glargine Combination With Exenatide Bid vs Switching Premix Human Insulin to Aspart30 in T2DM With Inadequate Glycaemic Control on Premixed Human Insulin and Metformin: a Randomized, Open, Parallel Trial
Brief Title: Efficacy and Safety of Basal Insulin Glargine Combination With Exenatide Bid vs Aspart30 in T2DM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xuefeng Yu, Director of Department of Endocrinology, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10352
Record Dates: First submitted 2015-06-02; First posted 2015-06-10 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: exenatide; glargine; aspart 30
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Exenatide; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- glargine + exenatide (Experimental): Type 2 diabetic patients with inadequate glycaemic control on premixed human insulin and metformin previously. After a 12-week run-in period , switching premix human insulin to glargine ( once-daily subcutaneous injection at bedtime) combination with exenatide (subcutaneous injection, twice-daily).
  Interventions: Drug: glargine + exenatide
- aspart 30 (Active Comparator): Type 2 diabetic patients with inadequate glycaemic control on premixed human insulin and metformin previously. After a 12-week run-in period , switching premix human insulin to aspart 30 ( subcutaneous injection, twice daily).
  Interventions: Drug: aspart 30

INTERVENTIONS:
Drug: glargine + exenatide — glargine ( once-daily subcutaneous injection at bedtime) combination with exenatide (subcutaneous injection, twice-daily)
  Arms: glargine + exenatide
Drug: aspart 30 — aspart 30 ( subcutaneous injection, twice daily)
  Arms: aspart 30

SUMMARY:
Efficacy and Safety of Basal Insulin Glargine Combination with Exenatide bid vs Switching Premix Human Insulin to Aspart30 in T2DM with Inadequate Glycaemic Control on Premixed Human Insulin and Metformin: a Randomized, Open, Parallel trial.

DETAILED DESCRIPTION:
This is a multicentre, open-label, randomized and parallel trial that will compare the efficacy and safety of basal insulin glargine combination with Exenatide bid vs. switching premix human insulin to aspart30 in type 2 diabetic patients with inadequate glycaemic control on premixed human insulin and metformin. Approximately 248 patients will be enrolled in the study from China and randomized in a 1:1 ratio to one of the 2 treatment arms: once-daily insulin glargine + twice-daily exenatide + metformin; or twice-daily aspart 30 + metformin.

Study treatment will continue for 24 weeks. The primary efficacy measure is the change in HbA1c at 24 weeks. The study consists of 3 periods: a 1-week screening (period A), a 12-week run-in period (period B) and a 24-week treatment period (period C).

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Type 2 diabetic patients receiving twice-daily premixed human insulin 30 therapy ≥ 30 U/d and metformin with maximum tolerated dosage (≤ 1500mg/d)
* HbA1c > 8.0 % and < 11.0 % (HbA1c > 7.0 % and < 10.0% at randomization)
* Men and women (non-pregnant and using a medically approved birth-control method) aged ≥ 18 and ≤ 70 years
* BMI ≥ 23 and ≤ 35 kg/m2

Exclusion Criteria:

* Type 1 diabetes or other specific types of diabetes
* Pregnancy, preparation for pregnancy, lactation and women of child-bearing age incapable of effective contraception methods
* Uncooperative subject because of various reasons
* Abnormal liver function, glutamic-pyruvic transaminase (ALT) and glutamic-oxaloacetic transaminase (AST) > twice the upper limits of normal
* Impairment of renal function, serum creatinine: ≥ 133mmol/L for female，≥ 135mmol/L for male
* Serious chronic gastrointestinal diseases
* Edema
* Serious heart diseases, such as cardiac insufficiency (level III or more according to NYHA), acute coronary syndrome and old myocardial infraction
* Blood pressure: Systolic blood pressure (SBP) ≥ 180mmHg and/or diastolic blood pressure (DBP) ≥ 110mmHg
* White blood count (WBC) < 4.0×109/L or platelet count (PLT) < 90×109/L，or definite anemia (Hb：< 120g/L for male, < 110g/L for female), or other hematological diseases
* Endocrine system diseases, such as hyperthyroidism and hypercortisolism
* Experimental drug allergy or frequent hypoglycemia
* Psychiatric disorders, drug or other substance abuse
* Diabetic ketoacidosis and hyperosmolar nonketotic coma requiring insulin therapy
* Stressful situations such as surgery, serious trauma and so on
* Chronic hypoxic diseases such as pulmonary emphysema and pulmonary heart disease
* Combined use of drugs effecting glucose metabolism such as glucocorticoid
* Tumor, especially bladder tumor and/or family history of bladder tumor and/or long-term hematuria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
the absolute change in HbA1c from baseline to 24-week endpoint of basal insulin glargine combination with exenatide bid vs. switching to aspart30 in type 2 diabetic patients inadequately controlled on premixed human insulin and metformin. | from baseline to 24-week endpoint

SECONDARY OUTCOMES:
Change in HbA1c from baseline to 12 weeks endpoint | from baseline to 12 weeks endpoint
The percentage of participants who achieved HbA1c ≤ 6.5% and < 7% | 12 weeks and 24 weeks
Fasting blood glucose | 12 weeks and 24 weeks
Daily insulin use | baseline, 12 weeks and 24 weeks
Change in body weight | from baseline to 12 and 24 weeks
The incidence and rate of hypoglycaemic events during the study | baseline, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and technology, Wuhan, Hubei, China